CLINICAL TRIAL: NCT04177667
Title: Body Mass Index and Age Correlate With Antioxidant Supplementation Effects on Sperm Quality: Post-hoc Analyses From a Double-blind Placebo-controlled Trial
Brief Title: Body Mass Index and Age Correlate With Antioxidant Supplementation Effects on Sperm Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Ettore De Berardinis, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PXP-001A
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind placebo controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proxeed arm (Active Comparator): Subjects received 2 packets per day for 6 months of supplement (1000 mg of L-carnitine, 725 mg of fumarate, 500 mg of acetyl-L-carnitine, 1000 mg of fructose, 50 mg of citric acid, 50 µg of selenium, 20 mg of coenzyme Q10, 90 mg of vitamin C, 10 mg of zinc, 200 µg of folic acid and 1.5 µg of vitamin B12)
  Interventions: Dietary Supplement: Proxeed
- Placebo arm (Placebo Comparator): Subjects received 2 packets per day for 6 months of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Proxeed — Treatment with dietary supplement for male infertility for Proxeed Arm
  Arms: Proxeed arm
Other: Placebo — Treatment with placebo for Placebo Arm
  Arms: Placebo arm

SUMMARY:
Spermatozoa are vulnerable to lack of energy and oxidative stress as a result of elevated levels of reactive oxygen species. Therefore, it is essential that appropriate nutrients are available during maturation.

This randomized, double-blind, placebo-controlled trial investigated the effect of 6 months supplementation with carnitines and other micronutrients on sperm quality in 104 subjects with oligo- and/or astheno- and/or teratozoospermia with or without varicocele. Semen analyses were done at the beginning and end of the treatment. In addition to main analyses, post-hoc analyses for age and body mass index (BMI) were carried out. Results were interpreted by dividing the population into two age and BMI classes.

ELIGIBILITY:
Inclusion Criteria:

* men with oligo- and/or astheno- and/or terato-zoospermia
* with or without varicocele
* men aged between 18 and 50 years
* men from couples with history of difficulty conceiving for more than 12 months

Exclusion Criteria:

* subjects with known hypersensitivity to any of the treatment compound
* history of undescended testes or cancer
* endocrine disorders
* history of post-pubertal mumps
* genitourinary surgery
* obstructive azoospermia or obstructive pathology of the urogenital system
* autoimmune disease
* cystic fibrosis
* history of taking any therapy affecting fertility within last 3 months
* excessive consumption of alcohol or regular use of illicit or "recreational" drugs
* positive serology for HIV
* subjects following any special diet
* any condition which in the opinion of the investigator might put the subject at risk by participation in this study and subjects involved in any other clinical trials

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of sperm concentration (millions/ml) on spermogram of infertile men | 6 months
  Efficacy of the therapy on sperm concentration (millions/ml) of subject affected by male infertility with or without varicocele. Parameters have been compared in accordance with body mass index and age.
Evaluation of sperm motility (%) on spermogram of infertile men | 6 months
  Efficacy of the therapy on sperm motility (%) of subject affected by male infertility with or without varicocele. Parameters have been compared in accordance with body mass index and age.
Evaluation of sperm normal morphology (%) on spermogram of infertile men | 6 months
  Efficacy of the therapy on sperm normal morphology (%) of subject affected by male infertility with or without varicocele. Parameters have been compared in accordance with body mass index and age.

SECONDARY OUTCOMES:
Evaluation of pregnancy rate (number) | 6 months
  Pregnancy rate is the number of pregnancies including live births, still births and therapeutic abortions

IPD SHARING:
Plan to Share IPD: Yes